CLINICAL TRIAL: NCT04639895
Title: Use of Personalized Virtual Reality and Paper-and-pencil Interventions as Complementary Tools in the Treatment of Alcohol Use Disorder: From Cognitive Rehabilitation to the Prevention of Relapses.
Brief Title: Cognitive Rehabilitation Through Personalized Virtual Reality and Paper-and-pencil Interventions in the Alcohol Use Disorder Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Collaborators: Instituto São João de Deus (Unknown)
Responsible Party: Principal Investigator, Sergi Bermúdez i Badia, Associate Professor at the University of Madeira and Senior Researcher at NOVA-LINCS, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/20
Record Dates: First submitted 2020-10-27; First posted 2020-11-23 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol Use Disorder; Cognitive Rehabilitation; Virtual Reality; Paper-and-Pencil Tasks
MeSH Terms: conditions — Alcoholism | interventions — Paper; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (Experimental): Standard treatment protocol and 12 sessions (30 minutes each) of personalized cognitive activities in a virtual city environment (Reh@City).
  Interventions: Procedure: Virtual Reality
- Paper and Pencil (Experimental): Standard treatment protocol and 12 sessions (30 minutes each) of personalized paper-and-pencil cognitive activities,using the Task Generator tool.
  Interventions: Procedure: Paper and Pencil
- Control Group (Active Comparator): The standard treatment protocol.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Virtual Reality — The Virtual Reality group will be involved in the Standard treatment protocol and will perform personalized activities of daily living in a virtual city environment (Reh@City).
  Arms: Virtual Reality
Procedure: Paper and Pencil — The paper and Pencil group will be involved in the Standard treatment protocol and will perform personalized cognitive paper-and-pencil tasks, using the Task Generator tool.
  Arms: Paper and Pencil
Procedure: Control Group — The standard treatment protocol.
  Arms: Control Group

SUMMARY:
Cognitive dysfunction is one of the different consequences of excessive alcohol consumption, affecting many domains associated with prefrontal and temporal lobes, such as attention, verbal fluency, and memory.

This study will explore the clinical impact of two cognitive rehabilitation tools to promote cognitive improvements of AUD individuals.

DETAILED DESCRIPTION:
Excessive consumption of alcohol affects many functions associated with the prefrontal and temporal lobes, including different executive functions, memory, and complex motor control. Among several treatments, the Transtheoretical Model, a multidisciplinary approach, is one of the most standardized. However, it lacks effective and innovative cognitive rehabilitation tools. In this study, two cognitive rehabilitation tools, already clinically validated for stroke patients, will be implemented to promote cognitive recovery of Alcohol Use Disorder (AUD) individuals under treatment in the Alcoholic Rehabilitation Center S. Ricardo Pampuri from Casa de Saúde S. João de Deus (Madeira, Portugal). Within a randomized controlled trial with 60 participants, this study intend to assess and compare the clinical effectiveness of both a paper-and-pencil tasks training and content equivalent virtual reality (VR) simulation of activities of daily living with time-matched standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of Centro de Alcoologia Ricardo Pampuri (with Alcohol use Disorder diagnosis)
* Education (able to read and write)
* Standard neuropharmacological protocol

Exclusion Criteria:

* Abuse of other substances
* Neurological and psychiatric pathology (present or past)
* Severe depressive symptoms as assessed by the Beck Depression Inventory
* Visual problems that can affect the performance of the tasks (hemianopsy, diplopia)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (Cognitive Screening). | Baseline, Post-intervention (4 weeks), 6-month and 12-month follow-up
  Change from baseline in the Montreal Cognitive Assessment
Frontal Assessment Battery (FAB- Executive functioning). | Baseline, Post-intervention (4 weeks), 6-month and 12-month follow-up
  Change from baseline in the Frontal Assessment Battery.
SF-36 Medical Outcomes Study 36 - Item Short - Form Health Survey | Baseline, Post-intervention (4 weeks), 6-month and 12-month follow-up
  Change from baseline in the SF-36

SECONDARY OUTCOMES:
Toulouse-Pieron (Attention). | Baseline, Post-intervention (4 weeks), 6-month and 12-month follow-up
  Change from baseline in the Toulouse-Pieron Cancellation Test.
Verbal Paired Associates (WMS-III) (Memory). | Baseline, Post-intervention (4 weeks), 6-month and 12-month follow-up
  Change from baseline in the Verbal Paired Associates (WMS-III)
Rey Complex Figure (Visuospatial skills and visual memory). | Baseline, Post-intervention (4 weeks), 6-month and 12-month follow-up
  Change from baseline in the Rey Complex Figure.
Symbol Search and Coding (WAIS III). | Baseline, Post-intervention (4 weeks), 6-month and 12-month follow-up]
  Change from baseline in the Symbol Search and Coding (WAIS III)
Letter-number sequencing (WAIS-III)- Working Memory | Baseline, Post-intervention (4 weeks), 6-month and 12-month follow-up]
  Change from baseline in the Letter-number sequencing (WAIS III)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto São João de Deus- CSSJD Funchal, Funchal, Portugal

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT04639895/Prot_ICF_000.pdf